CLINICAL TRIAL: NCT05724953
Title: Alexithymia Intervention for Suicide (ALEXIS)
Brief Title: Alexithymia Intervention for Suicide
Acronym: ALEXIS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4089-P
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Suicide; Schizophrenia; Bipolar Disorder; Post Traumatic Stress Disorder; Major Depressive Disorder
MeSH Terms: conditions — Suicide; Schizophrenia; Bipolar Disorder; Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will attend 8 weeks of blended psychoeducation and digital mHealth (mobile health) intervention using smartphones designed to target poor emotion awareness to reduce suicide risk in veterans with SMI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Affective Awareness (Experimental): Intervention involving psychoeducation and daily emotion awareness practices
  Interventions: Behavioral: Affective Awareness

INTERVENTIONS:
Behavioral: Affective Awareness — Intervention involving psychoeducation and daily emotion awareness practices

SUMMARY:
Suicide rates among Veterans with Serious Mental Illness (SMI) are intractably high, representing a serious public health concern and a critical target for interventions. Yet, at present available treatments offer modest benefits. Thus, there remains an urgent need to identify novel approaches to address suicide risk in this population. Previous reports have linked suicide risk with poor social functioning. Emerging evidence from basic affective neuroscience research has indicated that effective social functioning is contingent on intact emotion awareness. Consistent with these findings, individuals with SMI at risk of suicide display social functioning difficulties along with poor emotion awareness (i.e., alexithymia). Employing a proof-of-concept design, the aim of the present study is to test the feasibility and acceptability of a novel, blended psychoeducation and digital mHealth (mobile health) intervention with smartphones designed to target alexithymia and poor social functioning to reduce suicide risk in Veterans with SMI.

DETAILED DESCRIPTION:
Suicide rates among veterans with Serious Mental Illness (SMI) are intractably high. Yet, at present available treatments offer only minimal to limited benefits to ameliorate this risk, despite a VA-wide implementation of enriched suicide prevention services and the availability of a national suicide hotline. This dire state represents a serious public health concern and a critical target for interventions. In response to this state, the Rehabilitation Research & Development Service (RR&D)'s Behavioral Health & Social Reintegration Program has highlighted the need for development of suicide prevention interventions that enhance social reintegration, functional outcomes, and improve overall participation in society. Germane to social functioning, extensive evidence from basic affective neuroscience research indicates that effective social functioning requires intact emotion awareness. Specifically, emotions are posited to provide crucial information about the significance of social situations and help to guide potential actions to be taken to navigate such situations. Negative emotional experiences in particular have critical informational value in signaling the need to adjust one's current state or activity. As different emotions may call for the use of distinct response strategies, lack of or reduced awareness of experienced feelings may make it difficult for individuals to choose response strategies for dealing effectively with social situations, resulting in poor social functioning. Consistent with these findings, recent reports indicate alexithymia, a transdiagnostic clinical syndrome characterized by poor emotion awareness, to be highly prevalent among veteran and civilians with SMI, with a recent large systematic review and meta-analysis indicating alexithymia predicting suicide ideation and behavior. Relatedly, previous reports indicate alexithymia has a detrimental impact on treatment outcomes. Altogether, these findings suggest alexithymia may play a key role in impacting suicide risk and treatment response in Veterans. Yet, despite its pervasiveness, chronic presentation, link to SMI and poor social functioning, and impact on clinical outcomes, the putative impact of alexithymia on suicide risk has not been investigated in Veterans with SMI at risk of suicide. Building on these findings, the goal of this project is to test the feasibility and acceptability of a novel, blended psychoeducation and digital mHealth (mobile health) intervention designed to target alexithymia and poor social functioning to reduce suicide risk in Veterans with SMI. Employing a proof-of-concept design, 40 participants will attend weekly group psychoeducation sessions targeting emotion awareness and social functioning along with an innovative mHealth emotion awareness skill training via smartphone to reduce alexithymia, enhance social functioning, and reduce suicide risk. Results from the present study will provide comprehensive characterization of suicide risk among Veterans with SMI, provide preliminary acceptability and feasibility data, and will inform the development of a randomized clinical trial to test the efficacy of the intervention to ameliorate suicide risk in this population.

ELIGIBILITY:
Inclusion Criteria:

* a DSM-V diagnosis of PTSD
* bipolar disorder
* MDD
* schizophrenia
* at risk of suicide(Columbia Suicide Severity Rating Scale
* C-SSRS >=3 or a suicide attempt in the past 5 years)

  * limited emotion awareness (Toronto Alexithymia Scale; TAS-20 >=52)
  * can understand all the study's risks and benefits

Exclusion Criteria:

* have medical/neurological conditions that could interfere with study participation
* enrolled in another treatment study
* unable/unwilling to provide a verifiable contact for emergency purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) Change | Baseline, 6 weeks, 8 weeks.
  A semi-structured interview indexing suicide risk and related domains including ideation, severity, intensity, behavior, and lethality.
Toronto Alexithymia Scale (TAS-20) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing difficulty identifying, difficulty describing feelings, and externally oriented thinking.
Provision of Social Relations Scale (PSRS) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing relationship with family and friends.

SECONDARY OUTCOMES:
Emotion Granularity Index Change | Baseline, 6 weeks, 8 weeks.
  An smartphone-based index of emotion granularity based on reports of emotions during daily functioning.

OTHER OUTCOMES:
MIRECC-GAF Change | Baseline, 6 weeks, 8 weeks.
  A rater-based index of occupational and social functioning.
World Health Organization Quality of Life - Brief (WHOQOL-BREF) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing quality of life.
Emotion Regulation Questionnaire (ERQ) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing emotion regulation.
Beck Depression Inventory (BDI) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing depressed mood.
Beck Anxiety Inventory (BAI) Change | Baseline, 6 weeks, 8 weeks.
  A self-report scale indexing anxiety.
Structured Clinical Interview for DSM-V Axis I (SCID-I) | Baseline.
  A rater-based clinical interview used to establish psychiatric diagnoses.
Clinician-Administered PTSD Scale for DSM-V (CAPS-V) | Baseline.
  A rater-based clinical interview used to assess trauma.
Childhood Trauma Questionnaire (CTQ) | Baseline.
  A self-report scale indexing childhood trauma.
Emotion Recognition task (ER-40) | Baseline, 8 weeks
  A standardized task indexing accuracy of recognition of emotions via photos of faces
Loneliness (UCLA Loneliness Scale) | Baseline, 8 weeks
  A self-report measure indexing sense of loneliness.
Emodiment of Emotions (EmBody Task) | Baseline, 8 weeks
  A standardized task indexing embodiment of emotions

CONTACTS AND LOCATIONS:
Overall Officials: David Kimhy, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No